CLINICAL TRIAL: NCT01690845
Title: Molecular Adsorbent Recirculating System (MARS®) for the Treatment of Patients With Hypoxic Hepatitis - a Prospective Randomized Controlled Clinical Study
Brief Title: Molecular Adsorbent Recirculating System (MARS®) in Hypoxic Hepatitis
Acronym: MARS in HH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Valentin Fuhrmann, Associate Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10712010
Record Dates: First submitted 2012-09-16; First posted 2012-09-24 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Hypoxic Hepatitis; Ischemic Hepatitis; Shock Liver; Hypoxic Liver Injury; Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Patients with severe HH will be treated with standard medical therapy (i.e. vasopressor support with norepinephrine in refractory hypotension = RR mean < 65 mmHg, positive inotropic support with dobutamine if the central venous oxygen saturation < 70%, renal replacement therapy in case of severe metabolic acidosis and/or renal failure, antibiotic treatment in case of suspected or proven infection, mechanical ventilation in case of severe hypoxemia or hypercapnia and/or GCS <= 8.
- MARS-Group (Experimental): 20 patients will be allocated by randomization to the MARS arm. Additionally to standard medical therapy they will receive 4 MARS sessions on three consecutive days, MARS® therapy will be applied for at least 12 hours per session. Thereafter, MARS® treatment will be continued if the patient still has increasing aminotransferase levels, requires vasopressor support or suffers from cholestasis (defined as serum bilirubin levels > 5 mg/dL) for 3 sessions again. There will be a maximum of 7 MARS ® sessions per patient.
  Interventions: Device: MARS

INTERVENTIONS:
Device: MARS — Molecular adsorbent recirculating system (MARS®) can be used in patients with acute liver failure for bridging to liver transplantation. Studies reported that MARS® therapy improved the hemodynamic situation in patients with acute and acute on chronic liver failure. Several groups observed an increase in arterial pressure, systemic vascular resistance index, a decrease in portal pressure and improvement of renal blood flow. Furthermore, studies demonstrated that MARS therapy reduces ammonia levels and improves hepatic encephalopathy.
  Other Names: Molecular adsorbent recirculating system (MARS®)
  Arms: MARS-Group

SUMMARY:
Hypoxic hepatitis (HH) is reported to be the most frequent cause of elevated aminotransferase levels in hospital. Up to 10 % of critically ill patients develop HH during the course of their intensive care unit (ICU) stay. Occurrence of HH is a life threatening event and ICU-mortality is reported to be up to 60%. Early therapeutic intervention is of central prognostic importance in patients with HH to improve the hemodynamic impairment as early as possible, to reduce hyperammonemia and hepatic encephalopathy, to avoid progression of organ failure and to improve outcome. Studies reported that Molecular Adsorbent Recirculating System (MARS®) therapy improved the hemodynamic situation in patients with acute and acute on chronic liver failure. The study hypothesis is that MARS® therapy in critically ill patients with severe HH improves hepatic hemodynamics and function and consecutively the course of the disease. 40 patients with suffering of severe HH with aminotransferase levels > 40 times the upper limit of normal of more than 12 hours will be randomized 1:1 to MARS® therapy (n=20) or conventional therapy (n=20). 4 MARS®-sessions will be performed on three consecutive days, each for at least 12 hours. Treatment will be continued under special circumstances. The maximum duration of the treatment phase is 7 days. The primary endpoint is the difference of the indocyanine plasma disappearance rate at day 7. The expected duration of the study is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* presence of severe hypoxic hepatitis with aminotransferase levels > 40 times the upper limit of normal
* duration of hypoxic hepatitis more than 12 hours
* age >/= 18 years

Exclusion Criteria:

* age < 18 years
* pregnancy
* DNR - order
* liver cirrhosis
* Cardiopulmonary resuscitation with unknown neurological outcome and/or hypoxic brain damage
* Expected survival of less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
difference of the indocyanine plasma disappearance rate (ICG-PDR) | Days 1-7
  The primary endpoint will be the difference of the indocyanine plasma disappearance rate (ICG-PDR) at day 7. Only in case of major differences in baseline values of ICG-PDR we will use the change from baseline to day 7 of ICG-PDR (delta ICG-PDR) as outcome. Assuming normal distribution of ICG-PDR, we will formally test the null-hypothesis of no difference between intervention group and control using an independent sample t-test. The assumption of a normal distribution will be founded on visually inspecting a histogram and using the Shapiro Wilks test for normal distribution. If the assumption of normality does not hold data will be compared using the Mann-Whitney U-test. A p-level of < 0.05 will be considered statistically significant. Furthermore a linear random coefficient model will be used to incorporate daily measurements of ICG-PDR during the course of the study in terms of a repeated measures design.

SECONDARY OUTCOMES:
duration of vasopressor support | 1-28
ICU - length of stay | 1-28
hospital - length of stay | 1-90
7-day mortality | 7 days
28 day mortality | 28 days
number of organ failure on day 7 | 7 days
number of organ failure on day 28 | 28 days
markers of liver function | 1-28
  especially occurrence of jaundice (defined as total bilirubin levels > 3 mg/dL) will be documented
number of vasopressor free days | 28 days
systemic hemodynamics | 7 days
  systemic blood pressure, heart rate, cardiac index, central venous oxygen saturation, systemic vascular resistance index, global enddiastolic volume index, stroke volume variation, extravascular lung water index, pulse pressure variation, intrathoracic blood volume index, cardiac function index, central venous pressure
number of complications of HH | 1-28
  following complications will be encountered: cholestasis, secondary sclerosing cholangitis, hepatic encephalopathy grade 3 & 4, hypoglycemia, intraabdominal hypertension, new onset of infections, renal failure, hepatopulmonary syndrome
biomarkers | 0-28
  blood samples will be collected the assess markers of inflammation, markers of endothelial function, markers of cardiac function, markers of cholestasis, markers of liver cell necrosis etc
duration of mechanical ventilation | 1-28
necessity of renal replacement therapy | 1-28
duration of renal replacement therapy | 1-28
90 days mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Valentin Fuhrmann, Prof, Principal Investigator — Medical University Vienna
Locations (2):
- Medical University Vienna, Dpt. of Internal Medicine 3, Div. of Gastroenterology and Hepatology, Vienna, Vienna, Austria
- University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany